CLINICAL TRIAL: NCT03606993
Title: Cooking With Iron Ingots: Assessing Feasibility and Natural History Among Infants in Resource-limited Settings
Brief Title: Iron Fish for Dominican Republic (DR) Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Lucky Iron Fish (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-012988
Record Dates: First submitted 2018-07-10; First posted 2018-07-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia
Keywords: Iron-deficiency; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lucky Iron Fish™ (LIF) (Experimental): For Mother-infant dyads enrolled into the LIF arm, mother receives a cooking supplement: one ~ 200g iron ingot.
  Interventions: Other: Lucky Iron Fish (TM) - An iron ingot that is a Cooking supplement
- Enhanced standard of care (eSOC) (No Intervention): For mother-infant dyads in the eSOC arm, families are not provided iron supplementation (consistent with standard of care) but have additional visits and laboratory monitoring beyond well-child care (enhanced).

INTERVENTIONS:
Other: Lucky Iron Fish (TM) - An iron ingot that is a Cooking supplement — For Mother-infant dyads enrolled into the LIF arm, mother receives one ~ 200g iron ingot, instructions on use: add 2-3 drops of lemon juice to one-liter of water, place iron ingot in water, bring to boil for 10 minutes, remove iron fish from water and then use that water for cooking or drinking.
  Arms: Lucky Iron Fish™ (LIF)

SUMMARY:
This study evaluates the feasibility of cooking with an iron ingot, Lucky Iron Fish™ (LIF), and evaluate the natural history of hemoglobins and iron status among infants of families using this iron ingot in a population with a high prevalence of iron-deficiency anemia. Participants are mother-infant dyads, and are randomized to one of two arms: Lucky Iron Fish™or enhanced standard of care.

DETAILED DESCRIPTION:
Iron deficiency and iron-deficiency anemia contribute significantly to global pediatric morbidity, predominantly affecting women and preschool aged children in resource-limited settings. Iron-deficiency in infancy has been linked to neurodevelopmental delay.

Current methods of iron repletion and supplementation have proved inadequate. The Lucky Iron Fish™ is a iron ingot, the size of a small bar of soap, that is made of pure iron. When boiled, it releases bioavailable iron into water, which is then used for food preparation and/or drinking. Participants in the LIF arm are instructed to acidify the water with citrus juice (provided).

All participants are followed at the same intervals to complete questionnaires and study-related labs.

ELIGIBILITY:
Inclusion Criteria:

* Mother ≥ 18 years of age
* A newborn delivered at ≥ 35 weeks
* Infant Child followed by (or will be followed by) affiliated clinic (Niños Primeros en Salud [NPS]) OR Infant delivered at Angel Ponce, the local maternity hospital of Consuelo, Dominican Republic.
* Mother is Spanish speaking
* Mother permission is provided (informed consent)

Exclusion Criteria:

* Maternal history of Sickle Cell Disease (homozygous)
* Concurrent enrollment in related study of LIF on anemia of young children (CHOP study #16-012631).
* Inability to understand and speak Spanish
* Severe cognitive impairment or severe psychiatric disease which would prohibit the answering of study questions

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin over time | 6-months and 12-months
  Investigators will assess changes in hemoglobin within each study arm and compare hemolgobin levels between study arms (intervention vs. standard of care). Hemoglobin will be measured in grams per deciliter (g/dL) and measured at 6-months, and 12-months. If data is normally distributed, a paired/dependent t-test will be used, if non-normal, a non-parametric test like Wilcoxon's Matched pairs test will be used.

SECONDARY OUTCOMES:
Rates of refusal | 12-months
  Rates of refusal to participate in study measured as proportion of subjects refusing to enter study compared to total number approached.
Retention | 12-months
  Within each study arm (Iron ingot vs. Oral iron supplementation), will calculate proportion lost to follow-up. Number of subjects lost to follow up divided total number of subjects enrolled at study entry.
Adherence to iron ingot use | 12-months
  Using a questionnaire with several likert-scale questions, we will assess adherence to iron ingot use. Questions include "When was the last time you used the Fish", "how often do you use the fish for meal preparation", "how often do you use the fish to prepare water", "how long do you typically boil the fish". The answer to each question has between 4-5 possible ordinal responses which will be converted into numerical data (1,2,3,4,5) and cumulative scores will be created to assess degree of use/adherence.
Difference in microbiomes and microbiota | 12-months
  Using results from rectal swabs, the study will compare the microbiome and microbiota of infants receiving LIF+citus vs. eSOC
Difference in microbiomes and microbiota | 12-months
  Using results from nasopharyngeal swabs, the study will compare the microbiome and microbiota of infants receiving LIF+citus vs. eSOC

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lowenthal, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Ninos Primeros en Salud, Consuelo, San Pedro de Macorís, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKee SG, Close R, Lowenthal E. Evaluation of Iron Deficiency Anemia in a Pediatric Clinic in the Dominican Republic. Ann Glob Health. 2017 May-Aug;83(3-4):550-556. doi: 10.1016/j.aogh.2017.07.004. PMID 29221528